CLINICAL TRIAL: NCT06713577
Title: Clinical Study of a 3D Shaded Zirconia for Chairside CAD/CAM Restorations
Status: Enrolling by invitation | Type: Observational
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Other Study IDs: C-RE-24-018; HUM00263115 (Other: Medical School Institutional Review Board)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Dental Prosthesis Failure; Dental Prosthesis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Group 1 Crowns: 35 crowns delivered with a universal resin cement (Calibra Universal + by Dentsply Sirona).
  Interventions: Device: CEREC Cercon 4D
- Group 2 Onlays: 35 onlays delivered with selective enamel etch, bonding agent, and universal resin cement (Prime & Bond Active with Calibra Universal + by Dentsply Sirona).
  Interventions: Device: CEREC Cercon 4D
- Group 3 Fixed Partial Dentures (FPD): 12 Fixed Partial Dentures (FPD) delivered with a universal resin cement (Calibra Universal + by Dentsply Sirona).

INTERVENTIONS:
Device: CEREC Cercon 4D — One investigational medical device is a new generation of a full contour zirconia restorative material (CEREC Cercon 4D/Dentsply Sirona) for chairside computer assisted design/computer assisted machines (CAD/CAM) restorations. It has an internal core of 4 mol% (4Y) zirconia transitioning to an external layer of 4/5 mol% (4/5 Y) zirconia with a three-dimensional gradient of shade from an inner chromatic layer to an external translucent layer that replicates the natural structure and appearance of a tooth. It is indicated for crowns, bridges, veneers, inlays and onlays and implant crowns Clinical Study of a 3D Shaded Zirconia for Chairside CAD/CAM Restorations The other investigational medical devices are a universal bonding agent (Prime and Bond Active/Dentsply Sirona) and dual-cure, self-adhesive resin cement (Calibra Universal
  +/Dentsply Sirona). They are used in combination to deliver ceramic and zirconia restorations.
  Groups: Group 1 Crowns; Group 2 Onlays

SUMMARY:
This investigation will be a prospective, longitudinal clinical trial to study the clinical performance of a new monolithic, 3D shaded zirconia material for computer assisted design and computer assisted machining for chairside restorations. The restorations will be evaluated for a period of up to five years. The study is called Clinical Study of a 3D Shaded Zirconia for chairside computer assisted design and computer assisted machining (CAD/CAM) chairside restorations intended to be part of the validation plan and post market follow-up of the following products: CEREC Cercon 4D, Calibra Universal +, and Prime and Bond Active.

DETAILED DESCRIPTION:
The primary aim is:

▪ Evaluate the longitudinal clinical performance of 3D shaded zirconia onlays, crowns, and fixed partial denture (FPD) over five years of clinical service. The restorations will be evaluated with modified FDI criteria for maintaining their esthetic, functional and biological properties.

The secondary aims are:

* Evaluate the resistance to material chipping and fracture of reduced thickness zirconia chairside computer assisted design and computer assisted machining (CAD/CAM) onlays, crowns, and fixed partial dentures (FPDs).
* Evaluate the short-term post-operative sensitivity associated with cementation techniques using a self-adhesive, universal resin cement and a selective etch/universal bonding agent with a universal resin cement.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-75 years.
* Willing and able to sign and date the informed consent form and the HIPAA form.
* Onlays and Crowns: Each patient should have at least one carious lesion, defective restoration, or fractured portion of the tooth to be restored on a maxillary or mandibular premolar or molar tooth. Each lesion, fracture, or defective restoration should exhibit sufficient size or loss of tooth structure requiring an onlay or crown restoration. The tooth should have at least one opposing tooth in occlusion and one adjacent tooth with an intact proximal contact. No more than eight teeth that are endodontically treated and restorable with an onlay or crown may be included in the study. All remaining teeth in the study will test vital and be asymptomatic at the beginning of treatment. No more than two restorations will be placed per patient. If a patient presents with more than two acceptable teeth for the study, molar teeth will be included prior to premolar teeth.
* Fixed Partial Dentures (FPDs): Each patient should have at least one missing tooth, either anterior or posterior, that is appropriate for replacement with a fixed partial denture. Abutment teeth will have healthy periodontal status with at least a 1:1 crown:root ratio. The FPD should have at least two opposing teeth in occlusion and one adjacent tooth with an intact proximal contact. Both abutment teeth must be asymptomatic prior to treatment. Endodontically treated teeth will be acceptable for abutments if nonmetallic cores can be placed to retain the FPD. FPDs may include 3 or 4 teeth as indicated by the clinical situation but must be within the 43 mm span of the mill block to manufacture it as described later. The patient cohort should include a mix of non-endodontically as well as endodontically treated teeth.

Exclusion Criteria:

* Unlikely to be able to comply with clinical study procedures, according to Principal Investigator's (PIs) judgment.
* Subject is not willing to participate in the clinical study.
* Patients unable to return for the recall appointments for a period of 5 years.
* Severe non-compliance to the clinical study plan as judged by the PI and/or Dentsply Sirona.
* Involvement in the planning and conduct of the clinical study. Applies to both Dentsply Sirona personnel and personnel from the clinical study site.
* Sensitive teeth.
* Teeth diagnosed with symptoms of incomplete tooth fracture.
* Teeth with a history of direct or indirect pulp capping procedures.
* Patients with significant untreated dental disease to include periodontitis and/or rampant caries.
* Women who self-report that they are possibly pregnant, pregnant, or lactating, as elective dental treatment is not indicated at these times.
* Patients with a self-reported history of allergies to the materials to be used in the study including composite resin cements, provisional acrylics, or zirconia restorative materials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population will be selected from current patients of either gender and any ethnic background, under clinical treatment at the University of Michigan Dental Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2031-01-22 (Estimated); Study Completion 2031-11-22 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the longitudinal clinical performance of 3D shaded zirconia onlays, crowns and FPDs. | At the five year follow up
  The restorations will be evaluated according to the modified World Dental Federation notation (FDI) criteria for maintaining their esthetic functional and biological properties.

SECONDARY OUTCOMES:
Evaluation of the longitudinal clinical performance of 3D shaded zirconia onlays, crowns and FPDs. | At the 6 month, 1 year, 2 year, 3 year and 4 year follow up
  The restorations will be evaluated according to the modified World Dental Federation notation criteria (FDI) for maintaining their esthetic functional and biological properties.
Evaluation of the resistance of the material chipping and fracture of the reduce thickness zirconia CAD/CAM onlays, crowns and FPDs. | At the 6 month, 1 year, 2 year, 3 year and 4 year and 5 year follow up.
  The restorations will be evaluated according to the modified World Dental Federation notation (FDI) criteria for maintaining their esthetic functional and biological properties.
Evaluation of the short-term post operative sensitivity associated with cementation techniques using a self-adhesive, universal resin cement and a selective etch/universal bonding agent with a universal resin cement. | Once a week after base line up to four weeks or until patient is asymptomatic.
  A criterion-referenced rating scale will be used to measure sensitivity (Scores 1-4)
  Sensitivity:
  1. = No sensitivity is experienced at anytime
  2. = Slight sensitivity is experienced occasionally but it is not uncomfortable
  3. = Moderate sensitivity is experienced intermittently, and it is noticeably uncomfortable
  4. = Severe discomfort is noted routinely with cold or pressure stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Fasbinder, Principal Investigator — Clinical Professor of Dentistry, Department of Cardiology, Restorative Sciences, and Endodontics
Locations (1):
- Department of Cariology, Restorative Sciences, and Endodontics at School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No